CLINICAL TRIAL: NCT02707367
Title: Recovery Roadmap Phase II: A Collaborative Multimedia Tool for Person-Centered Recovery Planning
Brief Title: Recovery Roadmap Phase II Small Business Innovation Research Grant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R44MH100712-03 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-14 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Mental Disorders; Behavior Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Roadmap (RR) Wave 1 (Experimental): All participants, in both Wave 1 and Wave 2, will act as their own comparator in a randomized stepped wedge design. Data collection in Wave 1 will include two pre-tests and two post-tests, building in an observation period that is not present in Wave 2.
  Interventions: Behavioral: Recovery Roadmap (RR) Wave 1
- Recovery Roadmap (RR) Wave 2 (Experimental): All participants, in both Wave 1 and Wave 2, will act as their own comparator in a randomized stepped wedge design. Data collection in Wave 1 will include one pre-test and three post-tests.
  Interventions: Behavioral: Recovery Roadmap (RR) Wave 2

INTERVENTIONS:
Behavioral: Recovery Roadmap (RR) Wave 1 — A web-based tool that provides guidance for implementing Person-Centered Recovery Planning. There are 3 components:
  1. Online module for service providers: A self-paced online module with interactive exercises, audio/video case studies, self-assessment, handouts, and collaborative materials designed for use with clients.
  2. Online module for people in recovery: A self-paced online module with interactive exercises, case studies, self-assessment, informational handouts, and collaborative materials to be completed with providers.
  3. Coaching & Support Center: A multimedia resource for providers with online coaching, a community of practice, and a resource library.
  Arms: Recovery Roadmap (RR) Wave 1
Behavioral: Recovery Roadmap (RR) Wave 2 — A web-based tool that provides guidance for implementing Person-Centered Recovery Planning. There are 3 components:
  1. Online module for service providers: A self-paced online module with interactive exercises, audio/video case studies, self-assessment, handouts, and collaborative materials designed for use with clients.
  2. Online module for people in recovery: A self-paced online module with interactive exercises, case studies, self-assessment, informational handouts, and collaborative materials to be completed with providers.
  3. Coaching & Support Center: A multimedia resource for providers with online coaching, a community of practice, and a resource library.
  Arms: Recovery Roadmap (RR) Wave 2

SUMMARY:
Recovery Roadmap: A Collaborative Multimedia Tool for Person-Centered Recovery Planning is a highly interactive web-based tool that provides guidance for providers and people in recovery, and promotes widespread implementation of Person-Centered Recovery Planning (PCRP). The Recovery Roadmap prototype was developed and tested by the Center for Social Innovation (C4), in partnership with Yale University's Program for Recovery and Community Health (PRCH), under a Phase I Small Business Innovative Research (SBIR) grant funded by the National Institute of Mental Health (NIMH) (1R43MH100712). Phase II refined the prototype Roadmap to streamline content, provide additional handouts and exercises for providers and clients to complete together, expand the audio/video vignettes and case studies, and add interactive online coaching and support for providers. Phase II also involved a robust evaluation of the Roadmap, using a quasi-experimental design in a fully powered trial. Approximately 30 practitioners and 90 clients (two to three clients per practitioner) were recruited from a total of five Community Support Programs in Connecticut. The programs were randomly selected into one of two intervention waves (Wave 1 and Wave 2). Survey data for Wave 1 included a total of four surveys: a pre-observation period, post-observation/pre-intervention, a midpoint survey (after completion of online curriculum), and a post survey (after completion of the entire intervention, including coaching calls). Surveys for the Wave 2 study participants included a pre-intervention, midpoint, and post survey. Qualitative interviews were also completed with interviews with practitioners and and administrators/clinical supervisors in each agency. State level client administrative client data were also collected and analyzed. Data examined changes in knowledge related to PCRP, person centered planning practices, practitioner/client relationship, and overall feedback on the intervention. our team also conducted a social network analysis to examine any changes in the size and strength of their networks related to person centered planning before and after the intervention. This phase will culminate with the dissemination of findings and preparation for Phase III commercialization.

DETAILED DESCRIPTION:
Person-Centered Recovery Planning (PCRP; also referred to as Patient-Centered Care Planning) is a field-tested intervention designed to maximize consumer choice and ownership of the treatment and recovery process. In Phase I of Recovery Roadmap: A Collaborative Multimedia Tool for Person-Centered Recovery Planning, the research team developed a prototype online tool to train providers and persons in recovery to understand and implement PCRP. The tool provided in-depth information and included interactive components (e.g., videos, fillable forms, case studies) to prepare users to partner effectively. The tool was pilot tested in two sites (one received the Recovery Roadmap only; the other received the tool plus a two-day in-person training) to obtain feedback about the Roadmap and determine its impact. The purpose of this Phase II SBIR study is to expand the Recovery Roadmap and conduct a fully powered study to determine the tool's effectiveness in training providers and supporting people in recovery in the PCRP process.

This proposed Phase II study design:

We propose a randomized stepped wedge design in which we will recruit a total of 30 practitioners and 90 persons in recovery (PIRs), 3-4 from each participating practitioner. Per the power analysis, 90 PIRs will have enough power to show statistical significance. We will:

* Randomize the sample into two intervention waves, Wave 1 and Wave 2.
* Do a T1 assessment with all practitioners and PIRs and then immediately begin the first 2-month component of Wave 1 Recovery Roadmap Intervention, i.e., the 5-unit, online PCRP curriculum, with both PIRs and practitioners (for Wave 1, T1 will be a Baseline assessment; for Wave 2, T1 will be a Pre-Baseline assessment). Total of 3 months, including assessment and completion of the curriculum, while Wave 2 completes an observation period.
* Do a T2 assessment (practitioners and PIRs) with both waves and launch the first component of intervention with Wave 2 (RR on-line training units only) while Wave 1 launches the second component of the RR intervention, i.e., practitioners (only) receiving 3 months of twice monthly coaching calls and an on-line Community of Practice. The series of web-based technical assistance (coaching) sessions are designed to reinforce PCRP key principles and practices as taught in the Recovery Roadmap and to optimize practitioners' use of/benefit from the web-based Community of Practice (COP). Wave 2 will have a total of 3 months, including its Baseline assessment and completion of the online curriculum. Wave 1 will have a total of 4 months, including the mid-point assessment for PIRs and practitioners and completion of coaching calls and COP for practitioners.
* Do a T3 Assessment (practitioners and PIRs). This will be, for Wave 1, a post-intervention assessment for PIRs and practitioners. For Wave 2, it will include a mid-point intervention assessment for PIRs and practitioners, with Wave 2 immediately beginning a second component of the intervention (3 months of twice monthly coaching calls and an online COP for practitioners). The series of web-based technical assistance sessions are designed to reinforce PCRP key principles and practices as taught in the Recovery Roadmap and to optimize practitioners' use of/benefit from the web-based Community of Practice. Wave 1 will have a total of 3 months, including assessments and a 2-month observation period. Wave 2 will have a total of 4 months, including the mid-point assessment for PIRs and practitioners and completion of coaching calls and COP for practitioners.
* Do a T4 Assessment (practitioners and PIRs) after Wave 2 has completed the COP. This is post intervention for Wave 2 and follow-up for Wave 1.

Hypotheses (for Aims 1 and 2):

H1: Providers in the RR condition will show statistically significant improvements in PCRP knowledge, skills, and provider-client relationships.

H2: Clients served by providers in the RR condition will show statistically significant improvements in treatment engagement and progress toward goals.

H3: Providers with higher levels of connectivity with their peers online will report sustained PCRP practices, compared with those with lower connectivity.

ELIGIBILITY:
Inclusion Criteria:

Clients:

* Age of majority
* Receipt of mental health services within the participating program;
* Directly work with a provider participating in the study
* The ability to participate in the activities as determined by the client's clinical team
* Willing and able to engage in a six month PCRP intervention and participate in follow-up research activities (24 months total including follow up assessments).

Providers: Providers must meet the following inclusion criteria:

* Age of majority
* Directly work with clients willing to participate in the study;
* Have access to and basic navigation skills for using the Internet (for online coaching
* Work for a participating program
* Have a willingness to engage in a six-month PCRP intervention and participate in follow-up research activities (24 months total).

Administrators: Inclusion criteria for administrators participating in key informant semi-structured interviews include:

* Age of majority
* Being administrator of a program participating in the study or umbrella organization
* Have access to a computer to view tool components
* Knowledge about the market for this type of product for use in adult mental health. The team will develop a screening tool for administrators to ensure they meet basic criteria for the study.

Exclusion Criteria:

Clients:

* Non-English speakers
* Clients who are unable to participate in study activities (per clinical team determination) and individuals who are unable to understand the informed consent process (per the Quiz of Understanding for Informed Consent) will be excluded from the study.

Providers:

* Non-English speakers
* Providers who have prior experience with RR tools will be excluded from the study.

Administrators:

• Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Person-Centered Care Questionnaire | PreBaseline (pre-observation), Baseline (pre-intervention), Time 1 (upon completion of the 6 month intervention), Time 2 (6 month follow-up), Time 3 (12 month follow-up)
  Change in PCRP knowledge and skills using the Person-Centered Care Questionnaire (Provider Version) for providers and the Person-Centered Care Questionnaire (Person in Recovery (PIR) Version) for clients (Tondora & Miller, 2009). The provider and client/PIR versions allow providers and clients/PIR to respond to slightly different items, but each study participant will have one reported PCCQ value at each time point.

SECONDARY OUTCOMES:
Recovery Knowledge Inventory | PreBaseline (pre-observation), Baseline (pre-intervention), Time 1 (upon completion of the 6 month intervention), Time 2 (6 month follow-up), Time 3 (12 month follow-up)
  Change in provider participant knowledge and attitude data on four domains: roles and responsibilities in recovery, non-linearity of the recovery process, roles of self definition and peers in recovery, and expectations regarding recovery (Bedregal et al., 2006).
Recovery Markers Questionnaire | PreBaseline (pre-observation), Baseline (pre-intervention), Time 1 (upon completion of the 6 month intervention), Time 2 (6 month follow-up), Time 3 (12 month follow-up)
  Change in client progress toward recovery (Ridgeway & Press, 2004).
Helping Relationship Inventory | PreBaseline (pre-observation), Baseline (pre-intervention), Time 1 (upon completion of the 6 month intervention), Time 2 (6 month follow-up), Time 3 (12 month follow-up)
  Change in the relationship between the provider and client using the Helping Relationship Inventory-Worker for providers and the Helping Relationship Inventory-Client for clients (Poulin & Young, 1997). Provider and client versions allow participants to respond to slightly different Helping Relationship Inventory (HRI) items, but each study participant will have one reported HRI value at each time point.

OTHER OUTCOMES:
Change in Provider Online Sociometric Surveys | PreBaseline (pre-observation), Baseline (pre-intervention), and Time 1 (upon completion of the 6 month intervention)
  Online Sociometric Surveys will contribute to a mixed methods approach of mapping provider social networks and social connectivity.
Qualitative Change in Provider Social Connectivity | PreBaseline (pre-observation), Baseline (pre-intervention), and Time 1 (upon completion of the 6 month intervention)
  Semi-structured qualitative interviews will contribute to a mixed methods approach of mapping provider social networks and social connectivity.
Change in Provider Network Analytic Data | PreBaseline (pre-observation), Baseline (pre-intervention), and Time 1 (upon completion of the 6 month intervention)
  Social network analytics will contribute to a mixed methods approach of mapping provider social networks and social connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ferreira, Ph.D., Principal Investigator — Center for Social Innovation; Janis Tondora, PsyD., Principal Investigator — Yale University Program for Recovery and Community Health
Locations (1):
- Center for Social Innovation, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedregal LE, O'Connell M, Davidson L. The Recovery Knowledge Inventory: assessment of mental health staff knowledge and attitudes about recovery. Psychiatr Rehabil J. 2006 Fall;30(2):96-103. doi: 10.2975/30.2006.96.103. PMID 17076052
- [Background] Poulin J & Young T. Development of a helping relationship inventory for social work practice. Research on Social Work Practice 7: 463-489, 1997.
- [Background] Ridgway P & Press A. Assessing the recovery-orientation of your mental health program: A user's guide for the Recovery-Enhancing Environment scale (REE) (version 1). Lawrence, Kansas: University of Kansas, School of Social Welfare, Office of Mental Health Training and Research. 2004.
- [Background] Tondora J & Miller R. The PCCQ: Person-centered care questionnaire: A tool for supervision and quality monitoring. Yale Program for Recovery & Community Health: New Haven, CT. 2009.